CLINICAL TRIAL: NCT05153993
Title: Effect of Stretching on Visco-elastic Behaviour of the Fascia Plantaris in a Healthy Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/1215
Record Dates: First submitted 2018-07-04; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Fasciitis, Plantar; Stretch; Rehabilitation; Stiffness of Unspecified Foot, Not Elsewhere Classified
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretch fascia plantaris (Experimental)
  Interventions: Other: Fascia stretch
- Control group (No Intervention)

INTERVENTIONS:
Other: Fascia stretch — Stretch of the fascia plantaris during 3x30", 5x/week, 6 weeks
  Arms: Stretch fascia plantaris

SUMMARY:
RCT with two arms: (1) stretch fascia plantaris (6 weeks, n=30) (2) control (n=30); Outcome parameters: ROM ankle and first toe; visco-elastic behaviour of the fascia plantaris determined by means of myotonometry Study protocol: Outcome parameters were evaluated before and after the intervention/control with a 6 weeks interval. All participants were screened bilaterally and for the participants assigned to the intervention group stretching was only performed on the dominant side

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Lower extremity injury

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Visco-elastic behaviour using myotonometry | within 20 minutes before and after intervention
  By means of the MyotonPro device

SECONDARY OUTCOMES:
Range of Motion of ankle joint and first metatarsalphalangeal joint | within 20 minutes before and after intervention
  By means of goniometry

CONTACTS AND LOCATIONS:
Overall Officials: Roel De Ridder, Principal Investigator — University Ghent
Locations (1):
- Roel De Ridder, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No